CLINICAL TRIAL: NCT04087603
Title: Teen School-Night Sleep Extension: An Intervention Targeting the Circadian System
Brief Title: Teen Sleep Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie Crowley, Associate Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HL112756 (NIH)
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Sleep Disorders, Circadian Rhythm; Adolescent Behavior
Keywords: Circadian rhythms; Sleep; Adolescence
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Adolescent Behavior

STUDY DESIGN:
Masking Description: Group assignment is impossible to blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekend Morning Bright Light & Early Bedtime (Experimental): * Assigned a set sleep schedule for 2 weeks
  * Receives evening time management goals to help facilitate scheduled bedtime
  * Receives morning bright light from 2 light boxes (Phillips EnergyLights) on two weekend mornings.
  Interventions: Behavioral: Weekend Morning Bright Light & Early Bedtime
- Healthy Control (No Intervention): - Sleep as usual at home for 2 weeks

INTERVENTIONS:
Behavioral: Weekend Morning Bright Light & Early Bedtime
  Arms: Weekend Morning Bright Light & Early Bedtime

SUMMARY:
The objective of this project is to develop an effective, yet feasible strategy to extend school-night sleep duration of older adolescents.

DETAILED DESCRIPTION:
The investigators are developing and testing a feasible behavioral intervention to increase school-night sleep duration by shifting the circadian system earlier and providing a time management plan for after-school activities in youngsters between 14 and 17 years and enrolled in high school. This study tests morning bright light and a school-night time management plan to facilitate earlier bedtimes to increase sleep duration. Circadian phase, sleep, neurobehavioral functioning and mood are measured before and immediately after the 2-week intervention and compared to a control group. Long-term effectiveness, adherence, and acceptability are also examined in a 3-week extension study. These data will provide evidence-based treatment strategies for delayed and sleep-restricted adolescents, and acceptability of and adherence to the treatment in this age group.

ELIGIBILITY:
Inclusion Criteria:

* 14- 17 years; enrolled in high school; lives in or near Chicago, IL

Exclusion Criteria:

-

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2019-05-12 (Actual)

PRIMARY OUTCOMES:
Change in circadian phase | Saturday evening before and Saturday evening after the 2-week intervention
  A change in the timing of the circadian system is measured using the Dim Light Melatonin Onset (DLMO), the most reliable measure of circadian phase in humans. Salivary melatonin is measured every 30 minutes in dim light and assayed using standard commercially-available radioimmunoassay (RIA) kits. The time at which melatonin rises above a 4 pg/mL threshold is the DLMO. The DLMO is measured before starting the intervention ("baseline DLMO") and then again after completing the 2-week intervention ("final DLMO"). The primary outcome is DLMO phase shift (baseline DLMO - final DLMO).
Change in sleep duration | 2-week baseline period and 2-week intervention period
  Sleep duration is measured from a wrist actigraph (Actiwatch Spectrum) worn on the non-dominant wrist throughout the month-long study. For the first 2 weeks, participants sleep as usual at home (baseline). During the last two weeks, the experimental group shifts their bedtime earlier and the control group does not. The main outcome is the change in average sleep duration from baseline to intervention weeks.
Change in daytime sleepiness | Saturday before and Saturday after the 2-week intervention
  Daytime sleepiness is derived from the Stanford Sleepiness scale (1=Feeling active, vital, alert, or wide awake; 7= no longer fighting sleep, sleep onset soon; having dream-like thoughts) administered as part of the Automated Neuropsychological Assessment Metrics (ANAM). Participants complete the ANAM on the Saturday preceding the intervention period and again on a Saturday after the intervention is over. The ANAM is administered 3 times throughout the day.
Change in daytime vigilance/attention | Saturday before and Saturday after the 2-week intervention
  Vigilance/attention is derived from simple reaction time test administered as part of the Automated Neuropsychological Assessment Metrics (ANAM). Participants complete the ANAM on the Saturday preceding the intervention period and again on a Saturday after the intervention is over. The ANAM is administered 3 times throughout the day. Outcomes include number of lapses (responses < 500 ms) and median reaction time. Changes in the the number of lapses and median reaction times are the main outcomes.
Change in inhibitory control | Saturday before and Saturday after the 2-week intervention
  Participants complete executive tests from the Delis-Kaplan Executive Function System (D-KEFS) on the Saturday preceding the intervention period and again on a Saturday after the intervention is over. The D-KEFS is a battery of executive-function tests that assess a broad range of higher-level cognitive skills. Inhibitory control is derived from the D-KEFS Color-Word Interference Test. Changes in completion time on this test is the main outcome.
Change in cognitive processing | Saturday before and Saturday after the 2-week intervention
  Participants complete executive tests from the Delis-Kaplan Executive Function System (D-KEFS) on the Saturday preceding the intervention period and again on a Saturday after the intervention is over. The D-KEFS is a battery of executive-function tests that assess a broad range of higher-level cognitive skills. Cognitive processing and monitoring is derived from the Design Fluency test. Changes in completion time and changes in the number of errors are the main outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will share the research data in publications. The sample size from this study allows for publishing the raw de-identified data, either in a table within the main text of the publication or in an appendix. The necessary precautions will be taken to ensure data are not linked to individual participants.

REFERENCES:
- [Derived] Crowley SJ, Velez SL, Killen LG, Cvengros JA, Fogg LF, Eastman CI. Extending weeknight sleep of delayed adolescents using weekend morning bright light and evening time management. Sleep. 2023 Jan 11;46(1):zsac202. doi: 10.1093/sleep/zsac202. PMID 36006948

DOCUMENTS (1):
  • Informed Consent Form (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04087603/ICF_000.pdf